CLINICAL TRIAL: NCT03898739
Title: What is the Preferred Angle of Traction to Decompress Cervical Nerve Roots?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Farag Hanafy, Lecturer of Biomechanics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Traction decompression angle
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Cervical Radiculopathy
Keywords: Traction; Decompression angles
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: One independent variable with many levels.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients with cervical radiculopathy, caused by cervical paramedian disc protrusion at C5-C6 or C6-C7 levels will participate in the study. They will be assigned randomly into three equal groups; A, B and C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- traction therapy from neutral position (Active Comparator): Patients in this group will receive traction decompression from neutral neck position with rope angle (0°)
  Interventions: Other: Cervical Traction from different angles
- traction therapy from lateral bending (Active Comparator): patients will undergo traction decompression from (30°) lateral bending of the neck toward the non-affected side
  Interventions: Other: Cervical Traction from different angles
- traction from flexion with lateral bending and rotation (Active Comparator): patients will be treated with traction decompression from (15°) neck flexion, (30°) lateral bending toward non- affected side and (15°) rotation to the affected side.
  Interventions: Other: Cervical Traction from different angles

INTERVENTIONS:
Other: Cervical Traction from different angles — Intermittent traction will be applied, maximum force will be 16 kg, minimum force will be 12 kg, traction cycle of each minute consists of 20 seconds static traction at the maximum force then released down to the minimum force for 20 seconds then repeated for 20 seconds static traction. Traction session time will be 15 minutes, and the traction force will be increased progressively with speed (50%) of increment of force

SUMMARY:
The purpose of the study is to investigate the effect of different angles of decompression on the Flexor Carpi Radialis (FCR) H-Reflex in patients with cervical radiculopathy

DETAILED DESCRIPTION:
Cervical traction has long been defined as a distracting force that separate the cervical segments and relieve nerve roots compression. Yet, there is lack of knowledge that reports the effects of different traction decompression angles and determines the proper angle of pull among different angles of decompression system

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study if they have C5-C6 and C6-C7 paramedian disc protrusion manifested by unilateral symptoms in C6-C7 roots dermatome and myotomes of the upper extremities, second grade of disc bulge (2-3mm) which was detected from T2 axial view of MRI, and diagnosed as cervical disc protrusion (C5- C7) for at least three months.

Exclusion Criteria:

- Patients will be excluded from the study if they have upper cervical spine disc pathology, cord compression and upper motor neuron symptoms, curvature abnormalities of the neck including reversed curve (kyphotic) and deformities, cervical rib syndrome, double crush syndrome, diabetic neuropathy, text neck, short neck (churchill neck), marked facet joint, neuro-central joint arthropathic pathology, osteoporotic patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
The Flexor Carpi radialis H-reflex | Changes from Baseline to 6-weeks after treatment
  The peak-to-peak amplitudes of four FCR-HR traces will be measured and averaged for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Samiha H Hassan, Prof., Study Chair — Professor of Physical Therapy for Neurology, Department of Physical Therapy for Neuromuscular Disorder and its Surgery, Faculty of Physical Therapy, Cairo University.; Shaymaa M Abdelmeged, PhD, Study Director — Lecturer at Department of Physical Therapy for Neuromuscular Disorder and its Surgery, Faculty of Physical Therapy, Cairo University.; Salam M Elhafez, Prof., Study Chair — Professor and Head of Department of Biomechanics, Faculty of Physical Therapy, Cairo University, Egypt

REFERENCES:
- [Background] Khan RR, Awan WA, Rashid S, Masood T. A randomized controlled trial of intermittent Cervical Traction in sitting Vs. Supine position for the management of Cervical Radiculopathy. Pak J Med Sci. 2017 Nov-Dec;33(6):1333-1338. doi: 10.12669/pjms.336.13851. PMID 29492054
- [Background] Liu J, Ebraheim NA, Sanford CG Jr, Patil V, Elsamaloty H, Treuhaft K, Farrell S. Quantitative changes in the cervical neural foramen resulting from axial traction: in vivo imaging study. Spine J. 2008 Jul-Aug;8(4):619-23. doi: 10.1016/j.spinee.2007.04.016. Epub 2007 Jun 21. PMID 17697801